CLINICAL TRIAL: NCT00991770
Title: Effect of Massage Therapy on Preoperative Anxiety and Postoperative Pain in Cancer Patients Undergoing Port Implantation
Brief Title: Massage Therapy and Port-a-Catheter Insertion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Massage Therapy Foundation (Other)
Responsible Party: Principal Investigator, Jennifer Rosen, Assistant Professor of Medicine, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H27681
Record Dates: First submitted 2009-10-06; First posted 2009-10-08 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2011-12

CONDITIONS: Cancer; Anxiety; Pain; Surgery
Keywords: Discomfort; Port-a-Catheters; Complementary and Alternative Medicine; Massage
MeSH Terms: conditions — Neoplasms; Anxiety Disorders; Pain | interventions — Massage

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Massage Therapy (Experimental): Massage therapy provided by a certified Massage Therapist
  Interventions: Other: Massage Therapy
- Control (Active Comparator): Empathic support conversation
  Interventions: Other: Attention Control

INTERVENTIONS:
Other: Massage Therapy — Two 20 minute chair massages: one before surgery and one after
  Arms: Massage Therapy
Other: Attention Control — Two 20 minute sessions where the Massage Therapist will talk to the patient about how they are feeling, listen, and provide empathetic support.
  Arms: Control

SUMMARY:
The purpose of this study is to assess the feasibility and efficacy of massage therapy for reducing pre-operative anxiety and post-operative pain among predominantly low income minority cancer patients undergoing surgical placement of a Port-a-Catheter.

DETAILED DESCRIPTION:
Despite major advances in the understanding of cancer and its treatment, patients continue to suffer greatly. Massage is now included in the National Comprehensive Cancer Network guidelines for the treatment of refractory cancer pain (1), and many cancer patients are turning to massage and other complementary therapies to help alleviate both their psychological and physical symptoms. However, complementary therapies, such as massage, are often unaffordable or unavailable to predominantly low-income cancer patients at safety net hospitals like Boston Medical Center.

The vast majority of cancer patients receiving chemotherapy undergo implantation of a permanent central venous access device, often referred to as a port implantation or implanted port. Although the implanted port carries multiple benefits for ease of treatment, after the procedure patients often complain of headaches, muscle stiffness and neck and shoulder pain that lasts for several days. Pain medication is the only therapy commonly offered for this and is often inadequate (2). Furthermore, since this is often the first surgical procedure for cancer patients at the beginning of their treatment, they often have significant levels of pre-procedure anxiety (3,4). Safe, efficacious, and cost-effective interventions that can reduce the anxiety and pain related to port implantation are needed.

This pilot study will look at how feasible and effective massage therapy is in reducing pre-operative anxiety and post-operative pain among BMC patients already undergoing surgical placement of an implanted port.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be adults within one month of diagnosis with any form of cancer.
* Patients must be scheduled to undergo, but have not yet received, port implantation.
* Patients must have the ability to understand and sign a written informed consent.

Exclusion Criteria:

* Patients who are unable or unwilling to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-02; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of massage therapy for reducing pre-operative anxiety among predominantly low income minority cancer patients undergoing surgical placement of an implanted port. | Baseline (prior to first 20 min intervention) and post-intervention/pre-surgery
Efficacy of massage therapy for reducing post-operative pain among predominantly low income minority cancer patients undergoing surgical placement of an implanted port. | Post-surgery/pre-second 20 min intervention and post-surgery/post-second 20 min intervention
Feasibility of using massage therapy to reduce pre-operative anxiety and post-operative pain among predominantly low income minority cancer patients undergoing surgical placement of an implanted port. | Day of surgery

SECONDARY OUTCOMES:
Effects of massage on the duration of the surgical procedure | Time of surgery
Effect of massage on the amount of anesthesia used during the surgical procedure | Time of surgery
Related costs of providing massage therapy to patients undergoing port-a-cath implantation | Day of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E Rosen, MD, FACS, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center - Ambulatory Surgery, Boston, Massachusetts, United States

REFERENCES:
- [Background] Vardy J, Engelhardt K, Cox K, Jacquet J, McDade A, Boyer M, Beale P, Stockler M, Loneragan R, Dennien B, Waugh R, Clarke SJ. Long-term outcome of radiological-guided insertion of implanted central venous access port devices (CVAPD) for the delivery of chemotherapy in cancer patients: institutional experience and review of the literature. Br J Cancer. 2004 Sep 13;91(6):1045-9. doi: 10.1038/sj.bjc.6602082. PMID 15316563
- [Background] Bow EJ, Kilpatrick MG, Clinch JJ. Totally implantable venous access ports systems for patients receiving chemotherapy for solid tissue malignancies: A randomized controlled clinical trial examining the safety, efficacy, costs, and impact on quality of life. J Clin Oncol. 1999 Apr;17(4):1267. doi: 10.1200/JCO.1999.17.4.1267. PMID 10561188
- [Background] Silvestri V, Nerini L, Missio G, Masini M, Faggi S, Gori A, Panella M. Levels of anxiety and pain during chemotherapy with peripheral versus central vascular access: an experimental evaluation. J Vasc Access. 2004 Oct-Dec;5(4):147-53. doi: 10.1177/112972980400500403. PMID 16596558
- [Background] Benedetti C, Brock C, Cleeland C, Coyle N, Dube JE, Ferrell B, Hassenbusch S 3rd, Janjan NA, Lema MJ, Levy MH, Loscalzo MJ, Lynch M, Muir C, Oakes L, O'Neill A, Payne R, Syrjala KL, Urba S, Weinstein SM; National Comprehensive Cancer Network. NCCN Practice Guidelines for Cancer Pain. Oncology (Williston Park). 2000 Nov;14(11A):135-50. PMID 11195407